CLINICAL TRIAL: NCT03048825
Title: A 2x2 Factorial Randomized Controlled Trial of Colchicine and Spironolactone in Patients with Myocardial Infarction / SYNERGY Stent Registry - Organization to Assess Strategies for Ischemic Syndromes 9
Brief Title: Colchicine and Spironolactone in Patients with MI / SYNERGY Stent Registry
Acronym: CLEAR SYNERGY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Boston Scientific Corporation (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLSYN.1702; OASIS-9 (Other: Population Health Research Institute)
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: ST Elevation Myocardial Infarction; Non ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Colchicine; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-dummy masking of colchicine and spironolactone in 2x2 factorial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Colchicine + Spironolactone +/- SYNERGY Stent (Active Comparator): Colchicine 0.5 mg tablet + Spironolactone 25 mg tablet.
  Trial participants who receive a SYNERGY Bioabsorbable Polymer Drug-Eluting Stent during their index PCI for STEMI will be included in the embedded SYNERGY Stent Registry.
  Interventions: Drug: Colchicine; Drug: Spironolactone; Device: SYNERGY Bioabsorbable Polymer Drug-Eluting Stent
- Spironolactone +/- SYNERGY Stent (Active Comparator): Colchicine-placebo tablet + Spironolactone 25 mg tablet.
  Trial participants who receive a SYNERGY Bioabsorbable Polymer Drug-Eluting Stent during their index PCI for STEMI will be included in the embedded SYNERGY Stent Registry.
  Interventions: Drug: Spironolactone; Device: SYNERGY Bioabsorbable Polymer Drug-Eluting Stent; Drug: Colchicine-Placebo
- Colchicine +/- SYNERGY Stent (Active Comparator): Colchicine 0.5 mg tablet + Spironolactone-placebo tablet.
  Trial participants who receive a SYNERGY Bioabsorbable Polymer Drug-Eluting Stent during their index PCI for STEMI will be included in the embedded SYNERGY Stent Registry.
  Interventions: Drug: Colchicine; Device: SYNERGY Bioabsorbable Polymer Drug-Eluting Stent; Drug: Spironolactone-Placebo
- Placebo +/- SYNERGY Stent (Placebo Comparator): Colchicine-placebo tablet + Spironolactone-placebo tablet.
  Trial participants who receive a SYNERGY Bioabsorbable Polymer Drug-Eluting Stent during their index PCI for STEMI will be included in the embedded SYNERGY Stent Registry.
  Interventions: Device: SYNERGY Bioabsorbable Polymer Drug-Eluting Stent; Drug: Colchicine-Placebo; Drug: Spironolactone-Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5 mg once daily
  Arms: Colchicine + Spironolactone +/- SYNERGY Stent; Colchicine +/- SYNERGY Stent
Drug: Spironolactone — Spironolactone 25 mg once daily
  Arms: Colchicine + Spironolactone +/- SYNERGY Stent; Spironolactone +/- SYNERGY Stent
Device: SYNERGY Bioabsorbable Polymer Drug-Eluting Stent — Trial participants who receive a SYNERGY™ Bioabsorbable Polymer Drug-Eluting (everolimus) Stent during their index PCI for STEMI will be included in the SYNERGY Stent Registry.
Drug: Colchicine-Placebo — Matching Colchicine-placebo once daily
  Arms: Placebo +/- SYNERGY Stent; Spironolactone +/- SYNERGY Stent
Drug: Spironolactone-Placebo — Matching Spironolactone-Placebo once daily
  Arms: Colchicine +/- SYNERGY Stent; Placebo +/- SYNERGY Stent

SUMMARY:
The CLEAR SYNERGY trial will study the long term effects of treatments following PCI to treat myocardial infarction. These treatments address both the culprit artery (PCI with SYNERGY stent) as well as the non-culprit arteries (randomization to routine colchicine and spironolactone).

DETAILED DESCRIPTION:
This is a multicenter, international SYNERGY stent registry that is embedded within a randomized, blinded, double-dummy, 2x2 factorial design trial of colchicine versus placebo and spironolactone versus placebo in patients with myocardial infarction who have undergone primary percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

1. a) Patients with STEMI referred for PCI within 12 hours of symptom onset, have a culprit lesion amenable to stenting, and with planned SYNERGY stent implantation for SYNERGY registry

   OR

   b) Patients with STEMI referred for PCI within 48 hours of symptom onset, not prospectively enrolled in SYNERGY stent registry

   OR

   c) Patients with diagnosis of Non STEMI with ischemic symptoms and either Hs Troponin > or = 300x ULN or Troponin > or = 200x ULN who have undergone PCI with one of the following:

   i. LVEF< or =45% ii. Diabetes iii. Multivessel CAD defined as 50% stenosis in 2nd major epicardial vessel iv. Prior MI v. Age >60 years
2. Able to be enrolled/randomized within 72 hours of index PCI (however patients should be randomized as soon as possible after PCI)
3. Written informed consent

Exclusion Criteria:

1. Age ≤18 years
2. Pregnancy, breastfeeding, or women of childbearing potential who are not using an effective method of contraception
3. Any medical, geographic, or social factor making study participation impractical or precluding required follow-up
4. Systolic blood pressure <90 mm Hg
5. Active diarrhea
6. Known allergy or contraindication to everolimus, the SYNERGY stent or any of its components
7. Unable to receive dual antiplatelet therapy
8. Any contraindication or known intolerance to colchicine or spironolactone
9. Requirement for colchicine or mineralocorticoid antagonist for another indication
10. History of cirrhosis or current severe hepatic disease
11. Current or planned use of any of: cyclosporine, verapamil, HIV protease inhibitors, azole antifungals, or macrolide antibiotics
12. Creatinine clearance <30 mL/min/1.73 m2
13. Serum Potassium >5.0 meq/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7264 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | up to 1 year
  Major Adverse Cardiac Events (MACE) for SYNERGY Stent (defined as the composite of death, recurrent target vessel MI, stroke, or ischemia driven target vessel revascularization) compared to performance goal
Composite of cardiovascular death, recurrent myocardial infarction, stroke, or unplanned ischemia driven revascularization | through study completion, an estimated average of 3 years
  The first occurrence of cardiovascular death, recurrent myocardial infarction, stroke, or unplanned ischemia driven revascularization in the colchicine comparison
Total composite events of cardiovascular death or new or worsening heart failure (co-primary 1) | through study completion, an estimated average of 3 years
  Total composite of cardiovascular death or new or worsening heart failure in the spironolactone comparison (co-primary 1)
Composite of cardiovascular death, new or worsening heart failure, recurrent myocardial infarction, or stroke (co-primary 2) | through study completion, an estimated average of 3 years
  The first occurence of cardiovascular death, new or worsening heart failure, recurrent myocardial infarction, or stroke in the spironolactone comparison (co-primary 2)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit S Jolly, MD, Principal Investigator — Population Health Research Institute
Locations (109):
- United States (11):
  - Central Cardiology, Bakersfield, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Illinois, Chicago, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Community Hospital, Munster, Indiana
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - NYU Langone Medical Center, New York, New York
  - The Christ Hospital Lindner Research Center, Cincinnati, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
- Australia (6):
  - Bankstown-Lidcombe hospital, Bankstown, New South Wales
  - SWSLHD - Campbelltown, Campbelltown, New South Wales
  - SWSLHD - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Peninsula Health, Frankston, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (22):
  - University of Alberta Hospital, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - Fraser Clinical Trials, New Westminster, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - William Osler Health, Brampton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston Health Science Centre, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - York PCI Group Inc, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Niagara Health System, Saint Catharines, Ontario
  - Scarborough Cardiology Research Associates Inc., Scarborough Village, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie - ULAVAL, Québec, Quebec
  - CIUSSS de l'Estrie - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec
  - PVRI - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (4):
  - Czech Center University Hospital Brno, Brno
  - St. Anne´s University Hospital, Brno
  - Karlovarska krajska nemocnice a.s., Karlovy Vary
  - University Hospital Královské Vinohrady, Prague
- Egypt (9):
  - Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Kharga Specialized Hospital, New Cairo, Kharga
  - Fayoum General Hospital, Al Fayyum
  - Tamia Central Hospital, Al Fayyum
  - Alexandria University Hospital, Alexandria
  - Beni Suef University Hospital, Banī Suwayf
  - Nasser Institute for Research and Treatment, Cairo
  - National Heart Institute, Giza
  - Suez Canal University Hospital, Ismailia
- France (3):
  - Centre Hospitalier Universitaire de Caen, Caen, Calvados
  - Centre Hospitalier Universitaire de Nimes, Nîmes
  - Institut de Cardiologie de la Pitié-Salpêtrière, Paris
- Hungary (3):
  - University of Debrecen, Debrecen
  - Bács-Kiskun County Hospital, Kecskemét
  - University of Szeged, Szeged
- Nepal (3):
  - Chitwan Medical College Teaching Hospital, Bharatpur, Bagmati Province/ State 3
  - Shahid Gangalal National Heart Centre, Kathmandu, Maharajgung
  - Manmohan Cardiothoracic Vascular and Transplant Center, Kathmandu
- Netherlands (16):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - St. Jansdal Ziekenhuis, Harderwijk, Gelderland
  - Tergooi Hospital, Hilversum, North Holland
  - ZiekenhuisGroepTwente (ZGT), Almelo, Overijssel
  - Beatrixziekenhuis, Gorinchem, South Holland
  - Franciscus Gasthuis, Rotterdam, South Holland
  - Bernhoven Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Gelderse Vallei Ziekenhuis, Ede
  - Admiraal de Ruyter Hospital, Goes
  - Groene Hart Ziekenhuis Gouda, Gouda
  - Radboud UMC, Nijmegen
  - Haga Hospital, The Hague
- North Macedonia (3):
  - PHI Clinical Hospital "Dr. Trifun Panovski", Bitola
  - University Clinic of Cardiology, Skopje
  - Clinical Hospital Tetovo, Tetovo
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Institute for Cardiovascular Diseases Dedinje, Belgrade
  - University Medical Center Zvezdara, Belgrade
  - Institute of Cardiovascular Disease Vojvodina, Kamenitz
- Spain (10):
  - Hospital Son Espases, Palma, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Clínic Barcelona Hospital Universitario, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias
  - Germans Trias i Pujol University Hospital, Badalona
  - Hospital Universitario La Paz, Madrid
  - Hospital Álvaro Cunqueiro, Vigo
- Switzerland (2):
  - Hôpitaux Universitaires de Genève, Geneva
  - Luzerner Kantonsspital, Lucerne
- United Kingdom (13):
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth, Dorset (county)
  - Castle Hill Hospital, Cottingham, East Riding of Yorkshire (unitary Authority)
  - Brighton & Sussex University Hospital NHS Trust, Brighton, East Sussex (county)
  - Lister Hospital, Stevenage, Hertfordshire (county)
  - William Harvey Hospital -East Kent Hospitals University NHS Foundation Trust, Ashford, Kent (county)
  - Norfolk and Norwich University Hospital, Norwich, Norfolk (county)
  - Kettering General Hospital, Kettering, Northamptonshire (county)
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire (county)
  - Ashford & St Peter's Hospitals NHS Foundation Trust, Chertsey, Surrey (county)
  - Salisbury NHS Foundation Trust, Salisbury, Wiltshire (county)
  - St. George's Hospital NHS Foundation Trust, London
  - The James Cook University Hospital, Middlesbrough
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jolly SS, d'Entremont MA, Lee SF, Mian R, Tyrwhitt J, Kedev S, Montalescot G, Cornel JH, Stankovic G, Moreno R, Storey RF, Henry TD, Mehta SR, Bossard M, Kala P, Layland J, Zafirovska B, Devereaux PJ, Eikelboom J, Cairns JA, Shah B, Sheth T, Sharma SK, Tarhuni W, Conen D, Tawadros S, Lavi S, Yusuf S; CLEAR Investigators. Colchicine in Acute Myocardial Infarction. N Engl J Med. 2025 Feb 13;392(7):633-642. doi: 10.1056/NEJMoa2405922. Epub 2024 Nov 17. PMID 39555823
- [Derived] Jolly SS, d'Entremont MA, Pitt B, Lee SF, Mian R, Tyrwhitt J, Kedev S, Montalescot G, Cornel JH, Stankovic G, Moreno R, Storey RF, Henry TD, Mehta SR, Bossard M, Kala P, Bhindi R, Zafirovska B, Devereaux PJ, Eikelboom J, Cairns JA, Natarajan MK, Schwalm JD, Sharma SK, Tarhuni W, Conen D, Tawadros S, Lavi S, Asani V, Topic D, Cantor WJ, Bertrand OF, Pourdjabbar A, Yusuf S; CLEAR investigators; CLEAR Investigators. Routine Spironolactone in Acute Myocardial Infarction. N Engl J Med. 2025 Feb 13;392(7):643-652. doi: 10.1056/NEJMoa2405923. Epub 2024 Nov 17. PMID 39555814
- [Derived] d'Entremont MA, Lee SF, Mian R, Kedev S, Montalescot G, Cornel JH, Stankovic G, Moreno R, Storey RF, Henry TD, Skuriat E, Tyrwhitt J, Mehta SR, Devereaux PJ, Eikelboom J, Cairns JA, Pitt B, Jolly SS. Design and rationale of the CLEAR SYNERGY (OASIS 9) trial: A 2x2 factorial randomized controlled trial of colchicine versus placebo and spironolactone vs placebo in patients with myocardial infarction. Am Heart J. 2024 Sep;275:173-182. doi: 10.1016/j.ahj.2024.06.007. Epub 2024 Jun 25. PMID 38936755
- [Derived] Akl E, Sahami N, Labos C, Genest J, Zgheib A, Piazza N, Jolly S. Meta-Analysis of Randomized Trials: Efficacy and Safety of Colchicine for Secondary Prevention of Cardiovascular Disease. J Interv Cardiol. 2024 Mar 12;2024:8646351. doi: 10.1155/2024/8646351. eCollection 2024. PMID 38505729
- [Derived] Granger CB, Pocock SJ, Gersh BJ. The need for new clinical trials of old cardiovascular drugs. Nat Rev Cardiol. 2023 Feb;20(2):71-72. doi: 10.1038/s41569-022-00819-1. No abstract available. PMID 36526898
- [Derived] Bouabdallaoui N, Tardif JC. Colchicine in the Management of Acute and Chronic Coronary Artery Disease. Curr Cardiol Rep. 2021 Jul 16;23(9):120. doi: 10.1007/s11886-021-01560-w. PMID 34269908
- [Derived] Silvis MJM, Demkes EJ, Fiolet ATL, Dekker M, Bosch L, van Hout GPJ, Timmers L, de Kleijn DPV. Immunomodulation of the NLRP3 Inflammasome in Atherosclerosis, Coronary Artery Disease, and Acute Myocardial Infarction. J Cardiovasc Transl Res. 2021 Feb;14(1):23-34. doi: 10.1007/s12265-020-10049-w. Epub 2020 Jul 9. PMID 32648087